CLINICAL TRIAL: NCT00661414
Title: A Multi-Center, Open-Label, Single-Arm, Phase 1, Dose Escalation Study of ASONEP (Sonepcizumab/LT1009) Administered as a Single Agent Weekly to Subjects With Refractory Advanced Solid Tumors
Brief Title: Safety Study of ASONEP (Sonepcizumab/LT1009) to Treat Advanced Solid Tumors
Acronym: ASONEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lpath, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT1009-Onc-001
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Solid Tumors
Keywords: Cancer; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — sonepcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: ASONEP (sonepcizumab/LT1009) — ASONEP [sonepcizumab/LT1009] is supplied as a colorless,particulate-free, pH 6.5, sterile solution containing approximately 10 mg/mL or 20 mg/mL of drug.
  The candidate drug is intended for single intravenous (iv) use administered over 90 minutes on a weekly basis.

SUMMARY:
The purpose of this study is to determine the safety, tolerability and highest dose of ASONEP that can safely be administered to patients with cancer who are no longer being helped by standard treatments.

DETAILED DESCRIPTION:
ASONEP™ (sonepcizumab/LT1009) is a humanized monoclonal antibody that possesses anti-angiogenic and anti-tumor activity in animal models of human cancer. ASONEP™ binds sphingosine 1-phosphate (S1P), a bioactive lipid signaling molecule that possesses potent pro-growth effects.

Preclinical studies with ASONEP™ (sonepcizumab/LT1009) and LT1002 (murine homolog of LT1009), demonstrate the potential of an anti-S1P treatment to reduce tumor volumes and metastatic potential, likely as a result of inhibiting new blood vessel formation needed to support tumor growth.

Lpath is developing ASONEP™ (sonepcizumab/LT1009) for the following therapeutic indication:

ASONEP™ [parenteral sonepcizumab (LT1009) for the treatment of cancer] is indicated for use in combination with TBD cytotoxic agents and other anti-angiogenic agents as second-line therapy to treat patients with an unresectable, locally advanced, recurrent or metastatic TBD cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years old.
* Must have a confirmed diagnosis of solid tumor that has been refractory to prior therapy and for which no additional therapy of known benefit is available.
* Must have measurable or non-measurable disease as defined by RECIST guidelines.
* Be male or non-pregnant, non-lactating female. A negative pregnancy test within one week prior to the start of the study if a female of childbearing potential.
* Subjects and their partners with reproductive potential must agree to use an effective contraceptive method (as deemed by the Investigator) while the subject is on study treatment and for 30 days after the last treatment.
* Must have a life expectancy of at least 3 months.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Must not be receiving any concurrent anticancer therapy.
* At least 4 weeks must have elapsed between any prior systemic treatment for the cancer (6 weeks for mitomycin and nitrosourea) and first dose of treatment on this protocol; at least 4 weeks must have elapsed between any prior radiation treatment for the cancer or major surgical procedure and the first dose of treatment on this protocol; all acute and chronic toxicities from prior treatment must have recovered to ≤ grade 1. Subjects with prostate cancer on Lupron® will be allowed to continue their treatment.
* Must have physical integrity of the gastrointestinal tract.
* Must have adequate organ and immune function as indicated by the following laboratory values:

  * Serum creatinine <1.5 x ULN or
  * Estimated creatinine clearance >45mL/min,
  * Total Bilirubin <2.0mg/dL (<34.2umol/L),
  * AST (SGOT) & ALT (SGPT) <3 x ULN,
  * Lymphocytes >LLN,
  * White Blood Cells >3.2 x 10^9cells/L,
  * Absolute Granulocyte Count >1.5 x 10^9cells/L,
  * HG >9g/dl without transfusion,
  * Platelets >100,000/µl.
* Must understand, be able, willing and likely to fully comply with study procedures, including scheduled follow-up, and restrictions.
* The subject must give written signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines, before completing any study related procedures.

Exclusion Criteria:

* Clinical evidence of active CNS involvement by malignancy. Subjects whose brain metastases were treated with radiation more than 8 weeks prior to entry on the trial, off steroids for at least 4 weeks, and with no evidence of disease progression in the brain for a minimum of 8 weeks are eligible for the trial.
* Active and uncontrolled infection.
* Hematologic cancers.
* Any uncontrolled medical problems, unrelated to the malignancy, or of sufficient severity that in the opinion of the Investigator, impair a subject's ability to give informed consent or unacceptably reduce the safety of the proposed treatment.
* Neurological or psychiatric disorders that would interfere with consent or study follow-up.
* Known or suspected intolerance or hypersensitivity to the study materials or closely related compounds] or any of their stated ingredients.
* History of alcohol or other substance abuse within the last year.
* Concurrent use of steroids or other immune suppressive agent.
* Known positive test for HIV.
* Evidence of bowel obstruction because of the theoretical possibility of GI perforation with an anti-angiogenesis agent.
* Female subjects who are pregnant or lactating.
* Subjects who have previously been enrolled into this study and subsequently withdrawn.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety | Jan 2009

CONTACTS AND LOCATIONS:
Overall Officials: William Garland, PhD, Study Director — Lpath, Inc.
Locations (3):
- United States (3):
  - Premiere Oncology, Scottsdale, Arizona
  - Pacific Oncology, San Diego, California
  - Premiere Oncology, Santa Monica, California

REFERENCES:
- [Background] Visentin B, Vekich JA, Sibbald BJ, Cavalli AL, Moreno KM, Matteo RG, Garland WA, Lu Y, Yu S, Hall HS, Kundra V, Mills GB, Sabbadini RA. Validation of an anti-sphingosine-1-phosphate antibody as a potential therapeutic in reducing growth, invasion, and angiogenesis in multiple tumor lineages. Cancer Cell. 2006 Mar;9(3):225-38. doi: 10.1016/j.ccr.2006.02.023. PMID 16530706